CLINICAL TRIAL: NCT06785090
Title: Effects of Topical Bromfenac Solution on Macular Thickness in Cataract Patients Undergoing Phacoemulsification Surgery
Brief Title: Effects of Bromfenac on Macular Thickness After Phacoemulsification Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inas Abd (Other)
Responsible Party: Sponsor-Investigator, Inas Abd, Sponsor-Investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-Bromphaco-2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Cataract; Cystoid Macular Edema After Phacoemulsification
Keywords: cataract; phacoemulsification; cystoid macular edema
MeSH Terms: conditions — Cataract; Macular Edema | interventions — bromfenac; Moxifloxacin; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bromfenac Group (Experimental): Participants in this group will receive bromfenac 0.09% ophthalmic solution as part of their postoperative care regimen following cataract surgery.
  • Interventions: 0.09% bromfenac ophthalmic solution twice daily in addition to Moxifloxacin 0.5% ophthalmic drops every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs for six weeks
  Interventions: Drug: Bromfenac; Drug: Moxifloxacin 0.5% ophthalmic solution; Drug: Dexamethasone phosphate 0.1%
- Control Group (Active Comparator): : Participants in this group will receive the standard postoperative care regimen without bromfenac.
  • Interventions: Moxifloxacin 0.5% every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs for six weeks
  Interventions: Drug: Moxifloxacin 0.5% ophthalmic solution; Drug: Dexamethasone phosphate 0.1%

INTERVENTIONS:
Drug: Bromfenac — Bromfenac is a non-steroidal anti-inflammatory drug (NSAID) formulated as a 0.09% ophthalmic solution. It is administered to reduce inflammation and prevent cystoid macular edema (CME) following cataract surgery.
  Arms: Bromfenac Group
Drug: Moxifloxacin 0.5% ophthalmic solution — antibiotic, standard postoperative care regimen
Drug: Dexamethasone phosphate 0.1% — steroid, standard postoperative care regimen

SUMMARY:
The goal of this clinical trial is to learn if bromfenac ophthalmic solution can prevent cystoid macular edema (CME) and reduce macular thickness in patients undergoing phacoemulsification surgery for cataract removal. The main questions it aims to answer are:

Does bromfenac reduce the incidence of CME after cataract surgery? Does bromfenac effectively control macular thickness postoperatively compared to standard care? investigators will compare the effects of bromfenac ophthalmic solution to a control group receiving standard postoperative treatment to see if bromfenac provides additional benefits.

Participants will:

Use bromfenac ophthalmic solution as prescribed postoperatively. Attend follow-up visits for macular thickness measurements and assessments of eye health.

Undergo routine postoperative evaluations to monitor for adverse effects.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the effectiveness of bromfenac ophthalmic solution in preventing cystoid macular edema (CME) and reducing macular thickness in patients who have undergone cataract surgery using phacoemulsification. Cataract surgery, while generally safe, can sometimes lead to complications such as CME, a condition that causes swelling in the macula and may impair vision. Bromfenac, a non-steroidal anti-inflammatory drug (NSAID), is commonly used after cataract surgery to reduce inflammation and prevent such complications.

The main questions this study aims to answer are:

Can bromfenac ophthalmic solution effectively lower the risk of CME after cataract surgery? Does bromfenac help maintain or reduce macular thickness more effectively compared to standard postoperative care? Are there any significant side effects or risks associated with bromfenac use in this context? investigators will compare the outcomes of patients treated with bromfenac ophthalmic solution to those who receive standard postoperative treatment without bromfenac. This will help determine whether bromfenac provides superior protection against CME and better management of macular thickness.

Participant Involvement:

Participants will:

Use bromfenac ophthalmic solution as prescribed, Undergo detailed eye examinations, including macular thickness measurements, before surgery and during follow-up visits.

Be monitored for any side effects or adverse reactions to bromfenac during the study period.

Attend scheduled follow-up visits for assessments, which may include optical coherence tomography (OCT) imaging and visual acuity tests.

This study is focused on improving the understanding of bromfenac's role in postoperative eye care and helping optimize treatment protocols for cataract surgery patients to ensure better outcomes and prevent vision-related complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older.
* Patients diagnosed with cataracts.

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients with glaucoma, ocular hypertension, pseudo-exfoliation syndrome, or any optic nerve disease.
* Patients with ocular diseases that might influence macular thickness, such as:
* Age-related macular degeneration
* Epiretinal membrane
* History of uveitis
* Intraoperative complications
* Traumatic cases
* Patients who have undergone previous ocular surgery in the same eye, such as:
* Vitrectomy
* Intravitreal injection
* Retinal laser therapy
* Corneal surgery
* Patients who developed severe adverse effects from other drugs or had complications intraoperatively or postoperatively unrelated to bromfenac.
* Patients taking antiglaucoma medications.
* Patients lost to follow-up.
* Patients with an allergy to one of the postoperative medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid R Hussein, consultant ophthalmologist, Study Director — Ibn Al Haitham eye teaching hospital.
Locations (1):
- College of Medicine, University of Baghdad, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the plan to share individual participant data (IPD) is undecided. While the raw data from this study has been deposited in the public repository Zenodo to ensure accessibility, further decisions on sharing additional data or providing access to specific datasets will depend on future collaborations, publication requirements, and institutional guidelines.

REFERENCES:
- See also: This link provides access to the de-identified raw data from the clinical trial investigating the effects of bromfenac on macular thickness in cataract patients following phacoemulsification surgery. — https://doi.org/10.5281/zenodo.14318557
- Available data/document: Individual Participant Data Set: inas.abd2206m@comed.uobaghdad. — https://doi.org/10.5281/zenodo.14318557 — This link provides access to the de-identified raw data from the clinical trial investigating the effects of bromfenac on macular thickness in cataract patients following phacoemulsification surgery.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the outpatient clinic at Jenna Ophthalmic Center. Eligible patients were adults aged 40-75 years with cataracts undergoing phacoemulsification surgery. Recruitment was done through clinic referrals and patient consultations. Patients were informed about the study and consent was obtained before enrollment.
Pre-assignment Details: All participants underwent a pre-operative assessment, including eye exams, intraocular pressure measurements, visual acuity testing and a medical history review to screen for comorbidities. Eligible patients were randomized into two groups: Bromfenac treatment and control group.
Groups:
- Bromfenac Group: This group received Bromfenac 0.09% ophthalmic solution, applied twice daily for 6 weeks following phacoemulsification surgery. The treatment was aimed at preventing cystoid macular edema (CME) and reducing macular thickness post-operatively. Participants were monitored for efficacy and any adverse events during the follow-up period.
- Control Group: This group received Moxifloxacin 0.5% ophthalmic drops every 6 hours and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6 hours post-operatively, without administering Bromfenac 0.09% ophthalmic drops.
Period: Overall Study
Arm/Group | Bromfenac Group | Control Group
Started | 45 | 42
Completed | 45 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were reported for all participants enrolled in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac Group | Control Group | Total
Number analyzed (Participants) | 45 | 42 | 87
Sex: Female, Male [Count of Participants; unit: Participants] — The number and percentage of male and female participants in each group were recorded at baseline.
  Participants
    Female | 20 | 22 | 42
    Male | 25 | 20 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 24 | 43
  >=65 years | 26 | 18 | 44
Preoperative Macular Thickness [Mean (Standard Deviation); unit: Microns] — Mean central macular thickness (CMT) in microns (µm) before surgery, measured using optical coherence tomography (OCT).
  Microns | 252.6 (15.4) | 253.1 (14.8) | 252.8 (15.1)
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 45 | 42 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 42 | 87
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Adverse Events Related to Bromfenac
Description: This outcome evaluates the safety of bromfenac ophthalmic solution by assessing the incidence of adverse events related to its use after cataract surgery. Adverse events include corneal erosion, irritation, and any other complications recorded during follow-up visits up to 6 weeks postoperatively
Time Frame: 6 weeks postoperatively
Measure: Count of Participants; unit: Participants
Groups:
- Bromfenac Group: Participants who received bromfenac ophthalmic solution post-cataract surgery.
Arm/Group | Bromfenac Group
Number analyzed (Participants) | 45
Participants | 5

2. Primary Outcome: Change in Macular Thickness From Baseline to 6 Weeks Postoperatively After Cataract Surgery
Description: This outcome measures the change in macular thickness in participants treated with bromfenac ophthalmic solution compared to the control group. Macular thickness was assessed using Optical Coherence Tomography (OCT) at two time points: preoperatively (baseline) and 6 weeks postoperatively.
  The change was calculated as:
  Macular Thickness at 6 Weeks Postoperative - Baseline Macular Thickness. A negative value indicates a decrease (thinning), while a positive value indicates an increase (thickening) in macular thickness.
Time Frame: 6 weeks postoperatively
Population: All participants were included in the analysis, with no exclusions due to missing data, dropouts, or protocol violations
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Bromfenac Group | Control Group
Number analyzed (Participants) | 45 | 42
Microns | 252.6 (15.4) | 253.1 (14.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 6-week postoperative period following cataract surgery.
Description: Adverse events were defined as ocular complications during the 6-week postoperative period, including punctate epithelial erosion, ocular irritation, corneal edema, and intraocular pressure changes. Serious adverse events included significant visual impairment, infection, retinal detachment, or the need for surgery. Adverse events were assessed at follow-ups (1 day, 1 week, 6 weeks) through clinical exams, patient symptoms, and intraocular pressure measurements.
Groups:
- Bromfenac Group: Participants in this group will receive bromfenac 0.09% ophthalmic solution as part of their postoperative care regimen following cataract surgery.
  • Interventions: 0.09% bromfenac ophthalmic solution twice daily in addition to Moxifloxacin 0.5% ophthalmic drops every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs for six weeks
  Bromfenac: Bromfenac is a non-steroidal anti-inflammatory drug (NSAID) formulated as a 0.09% ophthalmic solution. It is administered to reduce inflammation and prevent cystoid macular edema (CME) following cataract surgery.
  Moxifloxacin 0.5% ophthalmic solution: antibiotic, standard postoperative care regimen
  Dexamethasone phosphate 0.1%: steroid, standard postoperative care regimen
- Control Group: : Participants in this group will receive the standard postoperative care regimen without bromfenac.
  • Interventions: Moxifloxacin 0.5% every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs for six weeks
  Moxifloxacin 0.5% ophthalmic solution: antibiotic, standard postoperative care regimen
  Dexamethasone phosphate 0.1%: steroid, standard postoperative care regimen
Arm/Group | Bromfenac Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/42
Other Adverse Events (participants affected / at risk) | 5/45 | 0/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Group (N=45) | Control Group (N=42)
Punctate Epithelial Erosion (PEE) (Eye disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
This study had a small sample size (45 in Bromfenac group, 42 in control), limiting statistical power. The short follow-up period of 6 weeks may not capture long-term effects. Results were based on a single-center study in Iraq, reducing generalizability. Adverse events were reported subjectively, which may have led to underreporting. Further studies with a larger sample size, extended follow-up, and diverse populations are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT06785090/Prot_SAP_000.pdf